CLINICAL TRIAL: NCT05200286
Title: A Phase I, Single-dose, Parallel Group Study to Assess the Pharmacokinetics of Olorofim in Subjects With Renal Impairment
Brief Title: A Phase I Study to Assess the Pharmacokinetics of Olorofim in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: F901318-01-17
Record Dates: First submitted 2022-01-18; First posted 2022-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Severe renal impairment (Experimental): 120 mg olorofim
  Interventions: Drug: Olorofim
- Normal renal function (Active Comparator): 120 mg olorofim
  Interventions: Drug: Olorofim

INTERVENTIONS:
Drug: Olorofim — Single oral dose
  Other Names: F901318

SUMMARY:
A single oral dose study to investigate the PK and safety of olorofim in subjects with severe renal impairment compared to subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 70 years of age inclusive, at the time of signing the informed consent.
* Body weight ≥50 kg and BMI within the range 18 to 35 kg/m2 (inclusive)
* Subjects with severe renal impairment (or End-Stage Renal Disease who are not on dialysis) and with an eGFR <30 mL/min, estimated using the Cockcroft-Gault equation at screening and Day -1
* Subjects with normal renal function must be in good health, as determined by a medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations
* Subjects with normal renal function are matched by gender, age (±10 years) and BMI (± 20%) to at least one renally impaired subject.

Exclusion Criteria:

* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study
* Subjects with any history of convulsion (other than childhood febrile convulsion before the age of 6 years).
* Subjects who have any clinically significant allergic disease (excluding mild or seasonal allergies such as contact dermatitis or hay fever) as determined by the Investigator.
* Subjects with a history of or any concomitant active malignancy.
* Subjects with a history of drug or alcohol abuse.
* Subjects with, or with a history of, any clinically significant neurological, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, ocular (including minor trauma), hematological, or other major disorders as determined by the Investigator.
* Subjects with signs or symptoms consistent with a COVID-19 infection at screening or Day -1
* Renally impaired subjects with kidney transplantation, or on dialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the time of the last quantifiable concentration (AUC 0-t) | 0-96 hours
Maximum Observed Plasma Concentration (Cmax) | 0-96 hours

SECONDARY OUTCOMES:
Time to Reach Maximum Plasma Concentration (Tmax) | 0-96 hours
Apparent Elimination Half Life (t1/2) | 0-96 hours
Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC 0-inf) | 0-96 hours
Number of Participants With Treatment-Emergent Adverse Events | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Omega Research, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No